CLINICAL TRIAL: NCT02206958
Title: Preventing Toileting Disability in Frail Older Women
Brief Title: Defeating Urinary Incontinence With Exercise Training (DUET) Feasibility Study
Acronym: DUET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1112S07944
Record Dates: First submitted 2014-07-30; First posted 2014-08-01 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Toileting Disability; Functional Urinary Incontinence
Keywords: Toileting disability; Functional urinary incontinence; Urinary incontinence; Frailty; Physical activity
MeSH Terms: conditions — Urinary Incontinence; Frailty; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No treatment control group (Other): No treatment control group
  Interventions: Behavioral: Defeating Urinary Incontinence with Exercise Training
- Behavioral Urinary Incontinence Treatment (Experimental): 12 week program combining behavioral treatments for urinary incontinence and physical activity
  Interventions: Behavioral: Defeating Urinary Incontinence with Exercise Training

INTERVENTIONS:
Behavioral: Defeating Urinary Incontinence with Exercise Training — 12 week multi-component program. Continence program administered by a nurse practitioner during 4 home visits. Participants do pelvic floor muscle exercises 5 days/week using a 13-minute instructional audio CD. Based on participant symptoms and preferences the following strategies are taught: bladder training, urge and suppression techniques, caffeine reduction, eliminating bladder irritants, medication adjustment, adequate fluid intake, constipation management, and reducing nocturia.
  2. Physical activity program including moderate intensity walking (30 minutes, 5 days weekly) and twice weekly group strength training sessions using Therabands led by a trained exercise instructor.

SUMMARY:
Pilot study to determine the feasibility and possible treatment effect of a multi-component intervention combining non-drug treatments for urinary incontinence and physical activity to improve urinary incontinence, toileting skills, physical function, and quality of life in frail older women without dementia living in senior housing facilities.

DETAILED DESCRIPTION:
This was a single blinded, two-arm pilot randomized controlled trial designed to test the feasibility and potential treatment effects of a multi-component intervention that combined behavioral urinary incontinence treatments with physical activity to improve urinary incontinence, toileting skills, quality of life, and physical function in frail older women without dementia living in senior apartment buildings.The intervention included a 12-week program of tailored behavioral UI treatments delivered by a nurse practitioner during 4 home visits, 150 minutes of weekly walking, and twice weekly strength training classes.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 60 years or older
* Have urinary incontinence
* Not currently meeting national recommendations for physical activity (150 minutes of weekly moderate intensity aerobic exercise and twice weekly strength building exercise.
* At risk for functional decline per the Vulnerable Elders Survey (score of 3+)
* Free of dementia (pass mini-cog screening)

Exclusion Criteria:

* Cognitive impairment
* Grade 4 vaginal prolapse or pessary use
* Orthopedic surgery in past year
* Urinary retention (catheter use)
* Neurological cause for urinary incontinence (i.e. Parkinson's Disease, MS)
* Bladder cancer
* Bladder or incontinence surgery in past year
* Recipient of hospice or palliative care
* Ostomy
* New prescription or dosage change in past three months for anti-incontinence medication

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Performance Oriented Timed Toileting Instrument (POTTI) | baseline, after completing 12 week intervention
  A performance based measure that takes less than 5 minutes to administer. Participants are timed as they complete tasks that simulate toileting including: rising from a chair, walking 15 feet to another chair, turning around, pulling down an elastic waist skirt worn over their typical clothing, sitting in the chair, grabbing a piece of toileting paper and throwing it into a wastebasket, rising and pulling the skirt back up. Longer times indicate greater difficulty with toileting. It has strong inter-rater and test-retest reliability (90% agreement) and has been validated with activities of daily living dependency (r= -.721, p<.001) in nursing home residents (Ouslander et al., 1987). It has demonstrated responsiveness to change in a recent clinical trial (van Houten et. al., 2007).
Toileting Skills Questionnaire | baseline, after completing 12 week intervention
  A five item toileting skills questionnaire that assesses participants level of difficulty with undressing, walking to the toilet, getting on and off the toilet, reaching to grab toilet paper, and reaching around to wipe their bottom. Responses for each item range from 0-no difficulty to 4-cannot do. Total scores range from 0-20. Higher scores indicate more difficulty.

SECONDARY OUTCOMES:
International Consultation on Incontinence Questionnaire (ICIQ) | baseline, after completing 12 week intervention
  A four item questionnaire reporting the frequency and amount of urine leakage, how much leakage interferes with everyday life, and when leaking occurs. Scores range from 0-21 with higher scores indicating greater severity.
3 day bladder diary | baseline, after completing 12 week intevention
Short Physical Performance Battery | baseline, after completing 12 week intervention
  Performance based test of balance, gait, and chair rising ability.
Environmental toileting barriers checklist | baseline
  Observation of environmental barriers to toilet access, i.e., inappropriate toilet seat height, grab bar placement, trip hazards on pathway to toilet, adequate lighting in bathroom and pathways to toilet and other barriers to easy toileting.
Incontinence Impact Questionnaire (IIQ) | baseline, after completing 12 week intervention
  The IIQ is a questionnaire with 30 items measuring the impact urinary incontinence has on social, physical, emotional, and psychological aspects of life. All items contain the same response options (0=not at all, 1=slightly, 2= moderately, 3=greatly) and scores range from 0-90.
Urogenital Distress Inventory (UDI) | baseline, after completing 12 week intevention
  The UDI has 20 items asking about how much urinary incontinence bothers the respondent. All items contain the same response options (0=not at all, 1=slightly, 2= moderately, 3=greatly) and scores range from 0-60.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota School of Nursing, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Talley KMC, Wyman JF, Bronas U, Olson-Kellogg BJ, McCarthy TC. Defeating Urinary Incontinence with Exercise Training: Results of a Pilot Study in Frail Older Women. J Am Geriatr Soc. 2017 Jun;65(6):1321-1327. doi: 10.1111/jgs.14798. Epub 2017 Mar 1. PMID 28248418